CLINICAL TRIAL: NCT00752141
Title: Cognitive Effects of Oral Oxybutynin and Oxybutynin Chloride Topical Gel in Older Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: OTG0801
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): oral oxybutynin
  Interventions: Drug: oxybutynin chloride immediate-release
- 2 (Experimental): oxybutynin topical gel
  Interventions: Drug: oxybutynin chloride topical gel
- 3 (Placebo Comparator): placebo tablets plus placebo gel
  Interventions: Other: placebo

INTERVENTIONS:
Drug: oxybutynin chloride immediate-release — capsule containing oxybutynin chloride immediate-release 5 mg tablet administered three times daily, and placebo gel administered once daily
  Arms: 1
Drug: oxybutynin chloride topical gel — oxybutynin chloride topical gel applied once daily, and capsule containing placebo tablet administered three times daily
  Arms: 2
Other: placebo — capsule containing placebo tablet administered three times daily, and placebo gel administered once daily
  Arms: 3

SUMMARY:
The purpose of this study is to explore the possible cognitive effects of oxybutynin tablets and oxybutynin gel.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 60 and over
* English as a primary language
* Given written informed consent by signing and dating an informed consent form prior to study entry

Exclusion Criteria:

* Current diseases in which the use of oxybutynin is contraindicated
* History of narrow-angle glaucoma or urinary or gastric retention
* Current use of drugs known to effect memory and cognition

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Measure of accuracy of delayed recall name-phase association test | one week

SECONDARY OUTCOMES:
Effects on other cognitive domains measured by various tests | one week

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tucson, Arizona
  - National City, California
  - Maitland, Florida
  - Naples, Florida
  - Ocala, Florida
  - Atlanta, Georgia

REFERENCES:
- [Derived] Kay GG, Staskin DR, MacDiarmid S, McIlwain M, Dahl NV. Cognitive effects of oxybutynin chloride topical gel in older healthy subjects: a 1-week, randomized, double-blind, placebo- and active-controlled study. Clin Drug Investig. 2012 Oct 1;32(10):707-14. doi: 10.1007/BF03261924. PMID 22909146